CLINICAL TRIAL: NCT06191341
Title: Consequences in ICU of Vaccination Status of Covid-19 Patients
Acronym: CIVIC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-11Obs-CHRMT
Record Dates: First submitted 2024-01-03; First posted 2024-01-05 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: SARS CoV 2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is a retrospective cohort study aiming to describe the characteristics, management and prognosis of vaccinated patients hospitalized in the intensive care unit (ICU), in comparison with non-vaccinated patients.

DETAILED DESCRIPTION:
In December 2019 started the first wave of Sars-Cov-2 virus infections in Wuhan, China : the start of a major, deadly global pandemic, which has so far caused more than 6 million deaths worldwide. In response to the scale of this pandemic, a large-scale vaccination campaign was rapidly in place, starting in December 2020. Despite this measure, admission of vaccinated patients to intensive care has been noticed. The aim of this study is to describe the characteristics, management and prognosis of vaccinated patients hospitalized in the intensive care unit (ICU), in comparison with non-vaccinated patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with Sars-Cov-2 pneumonia confirmed by positive reverse transcription polymerase chain reaction (RT-PCR) assay and hospitalized in the general intensive care unit of the CHR de Metz-Thionville, between 01/03/2020 and 01/06/2022.

Exclusion Criteria:

* missing data for primary or secondary outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with Sars-Cov-2 pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 1058 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
World Health Organisation (WHO) clinical progression scale | at hospital discharge
  highest score during hospital stay

SECONDARY OUTCOMES:
Mortality | at D28 after hospital admission
  Rate
Prognosis factors | at hospital admission
  Vaccinal status, SARS-COV2 variant, age, sex, BMI, SOFA score, hypertension, diabetus mellitus, immubodepression

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume LOUIS, MD, Principal Investigator — CHR Metz Thionville Hopital Mercy
Locations (1):
- CHR Metz-Thionville/Hopital Mercy, Metz, France

IPD SHARING:
Plan to Share IPD: No
According to the French law and the French Data Protection Authority (CNIL), we won't be able to publicly share individual participant data, but we plan to share their conclusions through peer-reviewed publications and conferences.